CLINICAL TRIAL: NCT00016523
Title: Inhaled Nitric Oxide for Preterm Infants With Severe Respiratory Failure
Acronym: Preemie iNO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Preliminary results showed increased intraventricular hemorrhage (IVH) in experimental arm
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Krisa P. Van Meurs, MD, Lead Principal Investigator, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICHD-NRN-0026; U10HD034216 (NIH); M01RR000032 (NIH); U10HD027904 (NIH); U10HD027853 (NIH); M01RR008084 (NIH); U10HD027856 (NIH); M01RR000750 (NIH); U10HD021397 (NIH); M01RR016587 (NIH); U10HD027880 (NIH); M01RR000070 (NIH); U10HD040689 (NIH); M01RR000633 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD027871 (NIH); M01RR006022 (NIH); U10HD040498 (NIH); M01RR007122 (NIH); U10HD040461 (NIH); U10HD040521 (NIH); M01RR000044 (NIH)
Record Dates: First submitted 2001-05-14; First posted 2001-05-16 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Respiratory Distress Syndrome (RDS); Sepsis; Pneumonia; Hypertension, Pulmonary
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Very Low Birth Weight (VLBW); Prematurity; Inhaled nitric oxide; Aspiration syndrome; Idiopathic pulmonary hypertension; Pulmonary hypoplasia
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome; Sepsis; Pneumonia; Hypertension, Pulmonary; Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled Nitric Oxide (Experimental): Inhaled Nitric Oxide
  Interventions: Drug: Inhaled nitric oxide
- Placebo (Active Comparator): Inhaled Oxygen
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inhaled nitric oxide — Started at 5 ppm and could be increased to 10 ppm
  Arms: Inhaled Nitric Oxide
Drug: Placebo — Started at 5 ppm and could be increased to 10 ppm
  Arms: Placebo

SUMMARY:
This multicenter trial tested whether inhaled nitric oxide would reduce death or the need for oxygen in preterm infants (less than 34 weeks gestational age) with severe lung disease.

DETAILED DESCRIPTION:
This multicenter, randomized, double-masked, controlled clinical trial evaluated the efficacy of inhaled nitric oxide (iNO) in the treatment of the preterm infant with respiratory failure secondary to respiratory distress syndrome (RDS), sepsis/pneumonia, aspiration syndrome, idiopathic pulmonary hypertension and/or suspected pulmonary hypoplasia.

Infants were followed until death or discharge to home. The trial compared iNO therapy to mock gas delivery as the control, and otherwise incorporated conventional management strategies (including treatment with surfactant and high frequency ventilation as adjuncts to iNO therapy).

During the initial dosing, iNO was started at 5 ppm and could be increased to 10 ppm. If the infant did not respond, study gas was discontinued. For infants who responded to study gas, a gradual weaning was initiated. The total exposure to study gas did not exceed 336 hours (14 days). Infants were monitored for signs of toxicity.

Medical and neurodevelopmental outcome of surviving infants were assessed at 18 to 22 months corrected age by masked, certified examiners.

ELIGIBILITY:
Inclusion Criteria

* Any infant with a birth weight 401 - 1500 grams and < 34 weeks gestational age with an OI (mean Paw x FiO2 x 100/PaO2) > 10 on two consecutive blood gases at least 30 minutes apart, but no more than 12 hours apart.

or

* Infants > 1500 grams and < 34 weeks gestational age will be entered in the Larger Preemie Pilot Study if they have an OI greater than or equal to 15 on two consecutive blood gases at least 30 minutes apart, but no more than 12 hours apart.
* Infants requiring assisted ventilation with a diagnosis of RDS/HMD, pneumonia and/or sepsis, aspiration syndrome, idiopathic pulmonary hypertension, or suspected pulmonary hypoplasia associated with PROM and/or oligohydramnios.
* Greater than or equal to 4 hours after one dose of surfactant.
* Less than or equal to 120 hours of age.
* All infants must have an indwelling arterial line.

Exclusion Criteria

* Any infant in whom a decision has been made not to provide full treatment (e.g. chromosomal anomalies or severe birth asphyxia).
* Known structural congenital heart disease, except patent ductus arteriosus and atrial-level shunts.
* Infants with any major abnormality involving the respiratory system such as congenital diaphragmatic hernia, tracheoesophageal fistula or cystic fibrosis.
* Any bleeding diathesis considered to be clinically significant or thrombocytopenia with platelet count < 50,000.
* Prior enrollment into a conflicting clinical trial such as the Neonatal Network Surfactant CPAP trial.Inclusion Criteria

Max Age: 120 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 420 (Actual)
Dates: Start 2001-01; Primary Completion 2003-09 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Death or Bronchopulmonary Dysplasia | At 36 weeks post-conceptional age

SECONDARY OUTCOMES:
Intraventricular Hemorrhage Grade III and IV | At 36 weeks post-conceptional age
Days on assisted ventilation | At 36 weeks post-conceptional age
Length of hospitalization | At hospital discharge
Retinopathy of prematurity | At hospital discharge
Air leaks | At 36 weeks post-conceptual age
Days on oxygen | At 36 weeks post-conceptual age
Supplemental oxygen | At 36 weeks post-conceptual age
Neurodevelopmental outcome | 18-22 months corrected age

CONTACTS AND LOCATIONS:
Overall Officials: Krisa P. Van Meurs, MD, Study Director — Stanford University; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Abbot R. Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Edward F. Donovan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; James A. Lemons, MD, Principal Investigator — Indiana University; Shahnaz Duara, MD, Principal Investigator — University of Miami; Charles R. Rosenfeld, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Jon E. Tyson, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University; T. Michael O'Shea, MD MPH, Principal Investigator — Wake Forest University; Neil N. Finer, MD, Principal Investigator — University of California, San Diego; Dale L. Phelps, MD, Principal Investigator — University of Rochester; Mark L. Hudak, MD, Principal Investigator — University of Florida; Robin H. Steinhorn, MD, Principal Investigator — Northwestern University; G. Ganesh Konduri, MD, Principal Investigator — Medical College of Wisconsin, Milwaukee
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - University of California at San Diego, San Diego, California
  - Yale University, New Haven, Connecticut
  - University of Florida, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Wayne State University, Detroit, Michigan
  - University of Rochester, Rochester, New York
  - Wake Forest University, Charlotte, North Carolina
  - RTI International, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Sokol GM, Ehrenkranz RA. Inhaled nitric oxide therapy in neonatal hypoxic respiratory failure: insights beyond primary outcomes. Semin Perinatol. 2003 Aug;27(4):311-9. doi: 10.1016/s0146-0005(03)00043-0. PMID 14510322
- [Result] Van Meurs KP, Wright LL, Ehrenkranz RA, Lemons JA, Ball MB, Poole WK, Perritt R, Higgins RD, Oh W, Hudak ML, Laptook AR, Shankaran S, Finer NN, Carlo WA, Kennedy KA, Fridriksson JH, Steinhorn RH, Sokol GM, Konduri GG, Aschner JL, Stoll BJ, D'Angio CT, Stevenson DK; Preemie Inhaled Nitric Oxide Study. Inhaled nitric oxide for premature infants with severe respiratory failure. N Engl J Med. 2005 Jul 7;353(1):13-22. doi: 10.1056/NEJMoa043927. PMID 16000352
- [Result] Van Meurs KP, Hintz SR, Ehrenkranz RA, Lemons JA, Ball MB, Poole WK, Perritt R, Das A, Higgins RD, Stevenson DK. Inhaled nitric oxide in infants >1500 g and <34 weeks gestation with severe respiratory failure. J Perinatol. 2007 Jun;27(6):347-52. doi: 10.1038/sj.jp.7211690. Epub 2007 Apr 19. PMID 17443204
- [Result] Hintz SR, Slovis T, Bulas D, Van Meurs KP, Perritt R, Stevenson DK, Poole WK, Das A, Higgins RD; NICHD Neonatal Research Network. Interobserver reliability and accuracy of cranial ultrasound scanning interpretation in premature infants. J Pediatr. 2007 Jun;150(6):592-6, 596.e1-5. doi: 10.1016/j.jpeds.2007.02.012. PMID 17517240
- [Result] Hintz SR, Van Meurs KP, Perritt R, Poole WK, Das A, Stevenson DK, Ehrenkranz RA, Lemons JA, Vohr BR, Heyne R, Childers DO, Peralta-Carcelen M, Dusick A, Johnson YR, Morris B, Dillard R, Vaucher Y, Steichen J, Adams-Chapman I, Konduri G, Myers GJ, de Ungria M, Tyson JE, Higgins RD; NICHD Neonatal Research Network. Neurodevelopmental outcomes of premature infants with severe respiratory failure enrolled in a randomized controlled trial of inhaled nitric oxide. J Pediatr. 2007 Jul;151(1):16-22, 22.e1-3. doi: 10.1016/j.jpeds.2007.03.017. PMID 17586184
- [Result] Ambalavanan N, Van Meurs KP, Perritt R, Carlo WA, Ehrenkranz RA, Stevenson DK, Lemons JA, Poole WK, Higgins RD; NICHD Neonatal Research Network, Bethesda, MD. Predictors of death or bronchopulmonary dysplasia in preterm infants with respiratory failure. J Perinatol. 2008 Jun;28(6):420-6. doi: 10.1038/jp.2008.18. Epub 2008 Mar 13. PMID 18337740
- [Result] Chock VY, Van Meurs KP, Hintz SR, Ehrenkranz RA, Lemons JA, Kendrick DE, Stevenson DK; NICHD Neonatal Research Network. Inhaled nitric oxide for preterm premature rupture of membranes, oligohydramnios, and pulmonary hypoplasia. Am J Perinatol. 2009 Apr;26(4):317-22. doi: 10.1055/s-0028-1104743. Epub 2008 Dec 9. PMID 19067285
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org